CLINICAL TRIAL: NCT05623813
Title: Individual- and Group-based Postoperative Education on Promoting Engagement in Daily Activities for Patients After Sternotomy: A Non-randomised Controlled Study
Brief Title: Individual- and Group-based Postoperative Education for Patients Sternotomy
Status: Completed | Type: Observational
Sponsor: University of Western Sydney (Other)
Collaborators: Liverpool Hospital (Unknown)
Responsible Party: Principal Investigator, Karen Liu, Prof, University of Western Sydney
Other Study IDs: UWesternSydney_Aug2022
Record Dates: First submitted 2022-11-01; First posted 2022-11-21 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Post-sternotomy
Keywords: patient education; individual and group delivery; engagement in daily activities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individual-based education: Participants in the individual-based education would receive tailored education on sternal precautions to facilitate engagement in daily activities.
  Interventions: Other: Postoperative education
- Group-based education: Participants in the group-based education would receive the same education on sternal precautions to facilitate engagement in daily activities.The group-based education included between two and five participants.
  They were invited to ask questions about their recovery and voice any concerns they had about being discharged home specific to their needs, covering a tailored portion of the education. Participants in group-based education had a chance to share their experiences and concerns with the group members.
  Interventions: Other: Postoperative education

INTERVENTIONS:
Other: Postoperative education — provide patients with the understanding and confidence to safely engage in their daily activities whilst following post-sternotomy precautionary guidelines throughout their recovery

SUMMARY:
Cardiac surgery via sternotomy is performed on more than one million people annually. Patient education may promote engagement in daily activities postoperatively. It is unknown if there is any difference in patients' feedback and outcomes when the education is delivered individually or in a group format.

The aim of this study is to collect participants' feedback and therapists' time spent on individual- and group-based Education in Daily Activities Engagement - Post-Sternotomy.

DETAILED DESCRIPTION:
This single-site non-randomised controlled study was conducted at Liverpool Hospital, NSW, Australia. All patients aged 18 or above who had received cardiac surgery via sternotomy at Liverpool Hospital cardiothoracic ward were consecutively allocated to the individual- or group-based postoperative education. Outcomes included a survey to obtain participants' feedback, the time spent by therapists delivering the education per participant, and participants' length of postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* had received cardiac surgery via sternotomy
* were medically ready for discharge

Exclusion Criteria:

* under the age of 18
* unable to provide consent
* did not speak English
* could not obtain a translator prior to discharge
* were infectious and required to isolate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 or above who had received cardiac surgery via sternotomy at Liverpool Hospital cardiothoracic ward.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Survey | Two to three days pre-discharge
  On participants' understanding, confidence, and satisfaction of the education
Survey | Four to six weeks post-discharge
  On participants' understanding, confidence, and satisfaction of the education

SECONDARY OUTCOMES:
Time spent delivering education per participant | Post-discharge, up to six weeks
  The time spent for each session was measured in minutes using a timer from the start to the end of the education delivery
Length of postoperative hospital stay | Post-discharge, up to six weeks
  Number of days between the date of surgery and the date of discharge

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not shared as per ethics protocol.